CLINICAL TRIAL: NCT02417740
Title: Natural History of Noncirrhotic Portal Hypertension
Status: Recruiting | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 150108; 15-DK-0108
Record Dates: First submitted 2015-04-15; First posted 2015-04-16 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01-12

CONDITIONS: Cystic Fibrosis; Immunologic Deficiency Syndrome; Turner Syndrome; Congenital Hepatic Fibrosis; Idiopathic Non-Cirrhotic Portal Hypertension
Keywords: Portal Hypertension; Portal Fibrosis; Liver Disease; Varices; Splenomegaly; Natural History
MeSH Terms: conditions — Cystic Fibrosis; Immunologic Deficiency Syndromes; Turner Syndrome; Hepatic Fibrosis, Congenital; Idiopathic Noncirrhotic Portal Hypertension; Hypertension, Portal; Liver Diseases; Varicose Veins; Splenomegaly

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Adult with absence of Portal Hypertension: Confirmed absence of Portal Hypertension will have no findings suggestive of non cirrhotic portal hypertension on liver biopsy and on portal pressure measurements on confirmatory examination.
- Adult with presence of Portal Hypertension: Confirmed Presence of Noncirrhotic Portal Hypertension, through confirmatory testing, tissue diagnosis by liver biopsy and/or portal hypertension (HVPG >5mmHg).
- Minors likely to have the absence of Portal Hypertension: Minors identified as Confirmed Absence of Noncirrhotic Portal Hypertension will have no abnormal findings on confirmatory examination.
- Minors likely to have the presence of Portal Hypertension: Minors identified as Confirmed Presence of Noncirrhotic Portal Hypertension, have shown they have the disease with a tissue diagnosis by liver biopsy and/or portal hypertension (HVPG >5).

SUMMARY:
Background:

- Noncirrhotic Portal Hypertension (NCPH) is caused by liver diseases that increase pressure in the blood vessels of the liver. It seems to start slowly and not have many warning signs. Many people may not even know that they have a liver disease. There are no specific treatments for NCPH.

Objectives:

- To learn more about how NCPH develops over time.

Eligibility:

- People age 12 and older who have NCPH or are at risk for getting it. In the past year, they cannot have had other types of liver disease that typically result in cirrhosis, liver cancer, or active substance abuse.

Design:

* Participants will have 2 screening visits.
* Visit 1: to see if they have or may develop NCPH.
* Medical history
* Physical exam
* Urine and stool studies
* Abdominal ultrasound
* Fibroscan. Sound waves measure liver stiffness.

<TAB>- Visit 2:

* Blood tests
* Abdominal MRI
* Echocardiogram
* Questionnaire
* Liver blood vessel pressure (hepatic venous portal gradient (HVPG)) measurement. This is done with a small tube inserted in a neck vein.
* They may have a liver biopsy.
* All participants will visit the clinic every 6 months for a history, physical exam, and blood tests. They will also repeat some of the screening tests yearly.
* Participants with NCPH will also have:
* Upper endoscopy test. A tube inserted in the mouth goes through the esophagus and stomach.
* At least every 2 years: Esophagogastroduodenoscopy.
* At least every 4 years: testing including HVPG measurements and liver biopsy.
* Participants without NCPH will also have:
* Liver biopsy and HVPG measurements to see if they have NCPH.
* Every 2 years: abdominal MRI and stool studies.
* The study will last indefinitely.

DETAILED DESCRIPTION:
Study Description:

Up to 400 subjects with noncirrhotic portal hypertension or at risk for developing noncirrhotic portal hypertension by virtue of their

underlying disease (as well as sporadic cases of noncirrhotic portal hypertension as referred to in this protocol) will be offered inclusion

in the study.

Objectives:

Primary Objective:

1. The goal of this natural history study is to generate understanding of the development and progression of NCPH. We will use our

findings to generate novel biomarkers that will enable improved follow-up of patients, assist in preventing complications, and

enhance transplant decision.

Secondary Objectives:

1. Measurement of the bile acids and lipids to understand NCPH and porto-systemic shunting.
2. Identification of the genetic modifiers of NCPH.
3. Evaluation of hepatic transcriptome in absence and presence of NCPH.
4. Characterization of microbiome signatures in NCPH.

Endpoints:

Primary Endpoints:

1. Establish surveillance methods and guidelines for evaluation of NCPH.
2. Develop an understanding of the biological mechanisms of the progression of NCPH.
3. Identification of novel biomarkers correlating with NCPH progression.

Secondary Endpoints:

1. Measurement of bile acids fractionated and total, as well as lipid panel to establish cut-off levels correlating with NCPH severity.
2. Establishment of positive or negative correlation between candidate susceptible genes and disease phenotype.
3. Identification of novel markers of fibrosis or the development of hepatic neoplasia from transcriptome analysis.
4. Characterization of microbiome signatures (taxonomic and functional), as well as identification of specific species.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Male or female, aged >= 18 years of age, and minors 12-17 years of age.
* Women of childbearing potential must agree to use birth control unless they are menopausal or had hysterectomy.
* Known diagnosis of NCPH, or to be at the risk for NCPH by virtue of underlying disease processes such as but not limited to; CGD, SCD, Mastocytosis, CVID, CF, and CHF.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnancy.
* Evidence of other forms of liver disease that typically result in cirrhosis.
* Evidence of active Chronic Hepatitis B infection as defined by the presence of hepatitis B surface antigen (HBsAg) in serum and elevated HBV DNA (>10,000 IU/mL).
* Hepatitis C as defined by the presence of hepatitis C RNA in serum.
* Evidence of other liver disease such as primary sclerosing cholangitis, primary biliary cirrhosis, Wilson s disease, autoimmune hepatitis as defined by either liver histology or laboratory abnormalities.
* Hemochromatosis as defined by presence of 3+ or 4+ stainable iron on liver biopsy or homozygosity for C282Y. Patients with iron saturation indices of >45% and serum ferritin levels of >300 ng/ml for men and >250 ng/ml for women will undergo genetic testing for hemochromatosis.
* Bile duct obstruction as suggested by imaging studies done within the previous six months.
* The presence of cirrhosis confirmed by liver biopsy.
* Active substance abuse, such as alcohol, inhaled or injection drugs within the previous one year (assessed during subject interviews by subject self-report).
* Evidence of hepatocellular carcinoma; either alpha-fetoprotein (AFP) levels greater than 50 ng/ml (normal <6.6ng/ml) and/or ultrasound (or other imaging study) demonstrating a mass suggestive of liver cancer.
* Evidence of cholangiocarcinoma as suggested by liver histology.
* Any other severe condition, which in the opinion of the investigators would impede the patient s participation or compliance in the study.
* Inability to comply or give written informed consent.

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with diagnosis of noncirrhotic portal hypertension above age of 12 years
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2015-07-27 (Actual); Primary Completion 2029-09-04 (Estimated); Study Completion 2029-09-04 (Estimated)

PRIMARY OUTCOMES:
To study the natural history of non cirrhotic portal hypertension. It is an ongoing study. | Ongoing
  natural history study

CONTACTS AND LOCATIONS:
Overall Officials: Theo Heller, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
This is a longitudinal study and it is not yet known if and when IPD will be made available.

REFERENCES:
- [Background] Sarin SK, Aggarwal SR. Idiopathic portal hypertension. Digestion. 1998 Jul-Aug;59(4):420-3. doi: 10.1159/000007502. No abstract available. PMID 9693222
- [Background] Sarin SK, Kumar A, Chawla YK, Baijal SS, Dhiman RK, Jafri W, Lesmana LA, Guha Mazumder D, Omata M, Qureshi H, Raza RM, Sahni P, Sakhuja P, Salih M, Santra A, Sharma BC, Sharma P, Shiha G, Sollano J; Members of the APASL Working Party on Portal Hypertension. Noncirrhotic portal fibrosis/idiopathic portal hypertension: APASL recommendations for diagnosis and treatment. Hepatol Int. 2007 Sep;1(3):398-413. doi: 10.1007/s12072-007-9010-9. Epub 2007 Sep 11. PMID 19669336
- [Background] Schouten JN, Garcia-Pagan JC, Valla DC, Janssen HL. Idiopathic noncirrhotic portal hypertension. Hepatology. 2011 Sep 2;54(3):1071-81. doi: 10.1002/hep.24422. Epub 2011 Jul 21. PMID 21574171
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-DK-0108.html